CLINICAL TRIAL: NCT03407677
Title: The Impact of ROTO Track® in Helping Patients With Diabetes Rotate Their Insulin Injections Better - a Proof-of-concept Study
Brief Title: The Impact of ROTO Track® in Helping Patients With Diabetes Rotate Their Insulin Injections Better
Acronym: ROTOone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peter Lommer (Other)
Responsible Party: Sponsor-Investigator, Peter Lommer, Head of Department, Endocrinology and Nephrology Department, Nordsjaellands Hospital
Organization: Nordsjaellands Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ROTOone
Record Dates: First submitted 2018-01-02; First posted 2018-01-23 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Diabetes
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Masking Description: During the baseline period patients will be blinded to the feature of the ROTO track®, which registers site of insulin injection and the features (vibration and light) that can assist the patient in rotation of injections. Patients will in the first week of the study be informed, that the ROTO track® is being developed as a new automatic device to register data on insulin injections including day, time and dose of insulin.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ROTO Track (Other): The individual patient will serve as his/her own control before intervention with ROTO Track
  Interventions: Device: ROTO track®

INTERVENTIONS:
Device: ROTO track® — An electronic injection form and injection log for keeping track of injection sites in the abdominal region. The device attaches directly to the insulin pen and activates whenever the insulin pen is picked up.

SUMMARY:
The ROTO track® is an electronic injection form and injection log for keeping track of injection sites in the abdominal region. The device attaches directly to the insulin pen and activates whenever the insulin pen is picked up. Small LED lights on the device will indicate where the next injection site is according to the individual patient's injection plan. By moving the pen and device to an "anchor point" in front of the navel, the device is able to start tracking where the insulin pen is being moved to. The device additionally contains a haptic interface to indicate to the user when the device has been moved to the next area in the injection plan.

The device registers the location, the time and the dosage automatically when the patient injects insulin with the pen

The rationale of the trial is that the ROTO track® can help patients rotate their injections sites and that this will provide the healthcare system with a new cost-effective tool for improving insulin injection techniques.

DETAILED DESCRIPTION:
Both observational and interventional studies have reported that proper rotation of injection sites can be obtained through intensive injection technique training, education and follow up of patients. Furthermore, this has significant beneficial effects on daily glycaemic variations, hypoglycaemic events, long term blood glucose levels, and insulin dose requirements. This is however frequently not done appropriately in every day practice.

At a small workshop at Nordsjællands Hospital in November 2017 with patients with type 1 diabetes the value of a device to registrar time, dose and rotation of insulin injections were discussed. All patients considered their own injection patterns as satisfying - although only one in four used a systematic approach. Most patients relied on their healthcare provider to identify side effects like lipohypertrophy, half of the patients re-used needles more than once and two took injections through the clothes now and then. All subjects would prefer a simple and small device to be used with the pen for the lifetime of the pen to minimize time used for injections and attraction of attention from other people.

The hypothesis is that the ROTO track® can reduce the number of insulin injections in the same subcutaneous skin area as compared with standard insulin injection instructions in patients with type 1 diabetes. The reduction of injection in same skin area will be quantified by a rotation score

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained before any trial related procedures are performed
2. Male or female aged 18 years
3. Type 1 diabetes with a duration of two or more years
4. Treated with three or more daily pen injections of Novo Rapid™ in the abdominal region
5. The subject must be willing and able to comply with trial protocol

Exclusion Criteria:

1. Blind or severely impaired eyesight
2. History of alcohol or drug abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-08-27 (Actual); Primary Completion 2019-11-20 (Actual); Study Completion 2019-11-27 (Actual)

PRIMARY OUTCOMES:
rotation of insulin injections | 6 days
  Number of insulin injections taken in a given subcutaneous skin area will be captured in a rotation score by the ROTO track® .
  The rotation score is a single ratio value that combines the distribution over the skin areas used with the time between re-use of a field. The value is set from 0 (meaning every injections in a single area) to 1 (meaning perfect rotation with the maximum possible time between two injections in the same skin area).

SECONDARY OUTCOMES:
rotation of insulin injections | 12 weeks
  Number of insulin injections taken in a given subcutaneous skin area captured in a rotation score by the ROTO Track
number of insulin infiltrates | 12 weeks
  documented by drawings and photos hereof
glucose variability | 12 weeks
  measured by continuous glucose monitors
glycaemic control | 12 weeks
  HbA1c
Insulin dose requirement | 12 weeks
  captured i diaries
Hypoglycaemic events | 12 weeks
  captured in diaries and by continuous glucose monitoring
Patient reported outcomes | 12 weeks
  quality of life
Patient reported outcomes | 12 weeks
  usability of the ROTO track®
Accuracy of the ROTO track® injection log | 12 weeks
  assessed by comparison of diaries and data from the ROTO Track

OTHER OUTCOMES:
Additional effect of an app in combination with the ROTO Track | Additional 12 weeks
  Number of insulin injections taken in a given subcutaneous skin area - captured in the rotation score
Insulin infiltrates - numbers | additional 12 weeks
  drawings documented by photography
Insulin dose requirement | additional 12 weeks
  from diaries
glycaemic control | additional 12 weeks
  measured by HbA1c

CONTACTS AND LOCATIONS:
Overall Officials: Peter L Kristensen, MD, PhD, Principal Investigator — Department of Clinical Research, Nordsjællands Hospital
Locations (1):
- Department of Clinical Research, Nordsjællands Hospital, Hillerød, Denmark